CLINICAL TRIAL: NCT04140162
Title: Phase 2 Study With Minimal Residual Disease (MRD) Driven Adaptive Strategy in Treatment for Newly Diagnosed Multiple Myeloma (MM) With Upfront Daratumumab-based Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2018.056; HUM00147751 (Other: University of Michigan)
Record Dates: First submitted 2019-10-21; First posted 2019-10-25 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Multiple Myeloma
Keywords: Dara-R; DaraRd; Dara-RVd; MRD
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Lenalidomide; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dara-Rd followed by Dara-RVd (Experimental): * Induction regimen with Daratumumab, Lenalidomide and Dexamethasone (Dara-Rd) in all study subjects, weeks 1-24
  * Consolidation regimen with Daratumumab, Lenalidomide, Bortezomib and Dexamethasone (Dara-RVd) in post-induction MRD+ population, weeks 25-36
  * Maintenance regimen with Daratumumab and Lenalidomide (Dara-R) in all study subjects, weeks 37-88
  * Maintenance regimen with lenalidomide (R) until progression or intolerance
  Interventions: Drug: Daratumumab; Drug: Lenalidomide; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab — Induction: 16 mg/kg actual body weight IV weekly (weeks 1-8; total of 8 doses) then every 2 weeks (weeks 9-24; total of 8 doses).
  Consolidation: 16 mg/kg actual body weight IV every four weeks (weeks 25-36)
  Maintenance: 16 mg/kg actual body weight IV every eight weeks (weeks 37-88)
  Sites will continue to use IV daratumumab to treat existing study patients until the IV daratumumab stock on site has been exhausted. The sites will then transition existing patient to SQ daratumumab. New patients will be started on SQ 1800mg daratumumab.
  Induction- Cycles 1-2 (days 1, 8,15, 22), Cycles 3-6 (Weeks 9-24- two weeks (days 1, 15 ) Consolidation- Every 4 weeks on day 1 Maintenance- Every 8 weeks on day 1
Drug: Lenalidomide — Induction: 25 mg PO once daily, on days 1-21 of each 28-day cycle (weeks 1-24)
  Consolidation: 25 mg PO once daily, on days 1-21 of each 28-day cycle (weeks 25-36)
  Maintenance: 10 mg PO once daily, on days 1-21 of each 28-day cycle until progression or intolerance
  Maintenance: 10 mg PO once daily, on days 1-21, weeks 37+ until progression
Drug: Bortezomib — Consolidation: 1.5 mg/m2 SQ on day 1, 8, 15 and 22 of each 28-day cycle (weeks 25-36)
Drug: Dexamethasone — Induction and Consolidation: 40 mg (or reduced dose of 20 mg) PO or IV weekly

SUMMARY:
This phase 2 trial will test whether the combination of DaraRd (daratumumab + lenalidomide + dexamethasone) as induction therapy, followed by DRVd (daratumumab + lenalidomide + bortezomib + dexamethasone) consolidation therapy, if needed, will result in more patients achieving minimal residual disease (MRD)-negative status, relative to the standard of care. Consolidation therapy will be administered only to those patients with MRD-positive status after induction therapy.

This is a study based on adaptive design for decision making of treatment options. Duration of therapy (daratumumab cycles) will depend on individual approach, response, evidence of disease progression and tolerance.

ELIGIBILITY:
INCLUSION

1. Participants ≥18 years of age or legal age of consent per local regulations (whichever is greater).
2. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.
3. ECOG status (Appendix A) of ≤2 and able to tolerate all applicable treatments per investigator's evaluation and standard institutional criteria.
4. Both transplant eligible and ineligible myeloma patients can be included in this study. If applicable, participant should be able to tolerate all treatments per investigator's evaluation, including high-dose chemotherapy and autologous stem cell transplant (ASCT) based on standard criteria at the institution where this treatment will be administered.
5. Participant must have a diagnosis of active MM according to International Myeloma Working Group (IMWG) diagnostic criteria.
6. Participant must also have measurable disease per protocol.
7. Baseline bone marrow or tissue sample available for Clonality ID in ClonoSEQ
8. Participant must be registered in and must comply with all requirements of REMSTM program for lenalidomide.
9. Female participant who:

   * Is post-menopausal for at least one year prior to study enrollment, OR
   * Is surgically sterile, OR
   * If of childbearing potential, must have a negative urine or serum pregnancy test within 10-14 days prior to and again within 24 hours of starting lenalidomide. They must also be willing to use TWO effective forms of contraception simultaneously from the time of signing the study consent until 90 days following the administration of the last dose of lenalidomide and 7 months following the administration of the last dose of bortezomib, OR
   * Agree to practice complete abstinence if that is aligned with their lifestyle, which does not include periodic abstinence or withdrawal.
10. Male participant, even if surgically sterilized, must agree to one of the following:

    * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of lenalidomide and 4 months following the administration of the last dose of bortezomib, OR
    * Agree to practice complete abstinence if that is aligned with their lifestyle, which does not include periodic abstinence or withdrawal.

EXCLUSION:

1. Diagnoses of smoldering MM (SMM), monoclonal gammopathy of undetermined significance (MGUS), non-secretory MM, plasma cell leukemia, AL amyloidosis, Waldenstrom's. macroglobulinemia, POEMS syndrome. History of SMM and/or MGUS is not excluded.
2. Known disease involvement of the CNS.
3. History of prior hematopoietic stem cell transplant of any type.
4. Received more than one cycle of anti-myeloma therapy prior to enrollment. Up to one cycle of myeloma therapy is allowed. Concomitant treatment is allowed with low-dose corticosteroids and bisphosphonates. The dose of corticosteroids for myeloma treatment should not exceed the equivalent of 160 mg of dexamethasone over a two-week period before initiation of protocol. Prednisone up to but no more than 10 mg po daily or its equivalent is allowed, for symptom management and comorbid conditions.
5. Significant renal insufficiency, defined as creatinine clearance <30ml/min per Cockcroft-Gault formula.
6. Hepatic impairment, defined as bilirubin >1.5 x institutional upper limit of normal (ULN) or AST (SGOT), ALT (SGPT), or alkaline phosphatase > 3x institutional ULN.
7. Absolute neutrophil count (ANC) < 1000 cells/mm3 within 14 days of enrollment. Growth factor may not be used to meet ANC eligibility criteria.
8. Hemoglobin (Hgb) < 8g/dL within 7 days of enrollment.
9. Platelet count < 75,000 cells/mm3 within 7 days of enrollment. Transfusion may not be used to meet platelet eligibility criteria.
10. Any condition, including laboratory abnormalities, that in the opinion of the investigator places the subject at unacceptable risk if subject were to participate in the study.
11. Major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from complications of the surgery.
12. Clinically significant peripheral neuropathy not well controlled with treatment, defined as symptoms limiting activities of daily living (basic ADLs).
13. Symptomatic uncontrolled cardiac disease including congestive heart failure with New York Heart Association class III-IV symptoms, arrhythmia, unstable angina or myocardial infarction within the past six months, or any other uncontrolled or severe cardiovascular condition.
14. Known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal.
15. Clinically uncontrolled asthma of any classification or known moderate or severe persistent asthma within the past two years (see asthma guidelines. https://www.nhlbi.nih.gov/files/docs/guidelines/asthma_qrg.pdf).
16. Serious intercurrent illness including but not limited to clinically relevant cerebrovascular disease, uncontrolled diabetes mellitus, cirrhosis, pulmonary disease.
17. Active autoimmune process or other disease requiring systemic immunosuppressive, monoclonal antibody, small molecule, or radiation therapy. However local radiation for myeloma related symptomatic treatment is allowed
18. Participant is:

    * Seropositive for HIV
    * Seropositive for Hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]
    * Subjects with resolved infection (i.e., subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded.
    * Participants with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
    * Seropositive for Hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy).
19. History of additional active malignancy in the past five years (not including squamous cell or basal cell carcinoma of the skin or in situ cervical cancer). However, malignancy treated with curative intent with <5% chance of disease relapse / recurrence in the next two years is allowed.
20. Known contraindication to study required medications (including steroids) or appropriate prophylactic medications (e.g. acyclovir, aspirin, warfarin or low-molecular weight heparin).
21. Women with a positive pregnancy test during the screening period prior to study initiation or who are lactating.
22. Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial.
23. Any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given.
24. Participants using strong CYP3A4 inducers are excluded unless the inducer can be switched to an alternative agent while receiving Bortezomib (per protocol).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2026-05-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who achieve MRD negativity either after induction or, if still MRD-positive after induction, after consolidation. | At the end of week 36 (post-consolidation therapy)
  Of participants who complete at least one cycle of induction therapy, proportion that achieve MRD-negativity after completion of induction + those who achieve MRD-negativity after completion of consolidation (if still MRD-positive after induction). MRD status determined by International Myeloma Working Group (IMWG) Response Criteria.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 3 years after start of study treatment
  Time from initiation of daratumumab-based combination regimen until death or last follow-up date (whichever occurs first).
Progression-free Survival (PFS) | Up to 3 years after start of study treatment
  Time from initiation of daratumumab-based combination regimen to disease progression, where disease progression is according to the IMWG criteria, death, or last disease evaluation before the start of any subsequent anti-myeloma therapy (whichever occurs first).
Proportion of participants who were MRD-positive after induction and subsequently achieve MRD-negative after consolidation. | At the end of week 36 (post-consolidation therapy)
  Of participants who are still MRD-positive after induction, proportion that achieve MRD-negative after consolidation. Per IMWG Response Criteria
Proportion of participants who maintain post-induction MRD-negativity to post-consolidation | At the end of week 36 (post-consolidation therapy)
  Of participants who achieve post-induction MRD-negativity, proportion that maintain MRD-negativity through completion of consolidation therapy.
Proportion of participants who maintain post-induction MRD-negativity to post-consolidation. | At the end of week 88 (post 1 year of maintenance therapy)
  Of participants who achieve post-induction MRD-negativity, proportion that maintain MRD-negativity through completion of 1 year of maintenance therapy.
Proportion of participants who maintain post-induction MRD-negativity to last follow-up visit. | After week 88, up to 3 years after start of study treatment
  Of participants who achieve post-induction MRD-negativity, proportion that maintain MRD-negativity until last follow-up visit (if after week 88).
Health-related quality of life assessment changes from baseline using EuroQol survey "EQ-5D." | Baseline to 16 weeks post-last-dose of study treatment (Dara, R, V or d)
  EQ-5D is a standardized participant-reported outcome measure developed by the EuroQol Group and used in this trial to assess health-related quality of life.
Neurotoxicity assessment changes from baseline using Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-Ntx) questionnaire. | Baseline to 16 weeks post-last-dose of study treatment (Dara, R, V or d)
  The FACT/GOG-Ntx is a patient-reported outcome measure used to assess health-related quality of life in patients undergoing cancer therapy, plus an eleven-item subscale (Ntx subscale) that evaluates symptoms and concerns associated specifically with chemotherapy-induced neuropathy.
Incidence of treatment-emergent adverse events | From start of study treatment (Dara-Rd) up to 30 days post last dose of study treatment (Dara, R, V or d)
  Toxicity will be assessed according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.
Proportion of participants with a successful stem cell mobilization after receiving Dara-based induction therapy. | At the end of week 24 (post-induction therapy)
  Of participants who have stem cells collected, proportion who have enough CD34+ cells after mobilization to be able to proceed with an autologous stem cell transplant (ASCT) if needed. Successful mobilization for each participant will be based on standard criteria at the institution where the transplant will be administered.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Ye, M.D., Study Director — MD Anderson
Locations (4):
- United States (4):
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Rochester, Rochester, New York
  - University of Texas Southwestern -- Simmons Comprehensive Cancer Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohan M, Gundarlapalli S, Szabo A, Yarlagadda N, Kakadia S, Konda M, Jillella A, Fnu A, Ogunsesan Y, Yarlagadda L, Thalambedu N, Munawar H, Graziutti M, Al Hadidi S, Alapat D, Thanendrarajan S, Zangari M, van Rhee F, Schinke C. Tandem autologous stem cell transplantation in patients with persistent bone marrow minimal residual disease after first transplantation in multiple myeloma. Am J Hematol. 2022 Jun 1;97(6):E195-E198. doi: 10.1002/ajh.26530. Epub 2022 Mar 21. No abstract available. PMID 35285981
- [Derived] Mohan M, Hari P, Szabo A, Dhakal B, Chhabra S, D'Souza A. Long term follow up of newly diagnosed multiple myeloma patients treated with pembrolizumab consolidation post-autologous stem cell transplantation. Leuk Res. 2021 Oct;109:106648. doi: 10.1016/j.leukres.2021.106648. Epub 2021 Jun 23. No abstract available. PMID 34182226